CLINICAL TRIAL: NCT03682237
Title: Optimizing Metabolic Control in Type 1 Diabetes With Multiple Daily Insulin Injections - Flash Glucose Monitoring, Carbohydrate Counting With Automated Bolus Calculation, or Both?
Brief Title: Optimizing Metabolic Control in Type 1 Diabetes - The Automatic Bolus Calculator Flash Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Hillerod Hospital, Denmark (Other); Hvidovre University Hospital (Other); Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other); Frederiksberg University Hospital (Other); Amager Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Nørgaard, Principal Investigator, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17040573
Record Dates: First submitted 2018-09-13; First posted 2018-09-24 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Hyperglycemia; Hypoglycemia; Carbohydrate counting; Automated bolus calculation; Flash glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A) Standard diabetes training (control) (No Intervention): More specifically, group training in general diabetes health issues, how to do experienced based dosing, how to handle sick days, exercise etc. in general terms. The group will not be taught in carbohydrate counting or bolus calculation. They will be encouraged to measure SMBG at least 4 times daily with patients own preferred glucose meter.
  Patients will be offered 6 months treatment with FGM after study end.
- B) Carbohydrate counting, automated bolus calculation (Active Comparator)
  Interventions: Device: Carbohydrate counting, automated bolus calculation
- C) Flash glucose monitoring (FGM) (Active Comparator): Group training with same content as for group A.
  Interventions: Device: Flash glucose monitoring (FGM)
- D) Carbohydrate counting, automated bolus calculation, FGM (Active Comparator): Group training as group B. A more sophisticated education concept will be developed for how FGM should be used to adjust settings and suggestions from the automated bolus calculator (MySugr app).
  Interventions: Device: Carbohydrate counting, automated bolus calculation; Device: Flash glucose monitoring (FGM)

INTERVENTIONS:
Device: Carbohydrate counting, automated bolus calculation — Group training in carbohydrate counting and bolus calculation. The app MySugr will be taught and downloaded on own smart phone and person specific parameters will be estimated and entered in the app with the patients. SMBG measures at least 4 times daily with patients own preferred glucose meter.
  Arms: B) Carbohydrate counting, automated bolus calculation; D) Carbohydrate counting, automated bolus calculation, FGM
Device: Flash glucose monitoring (FGM) — Group training, patients will be instructed to use unblinded FGM for the whole study period. Patients are recommended to measure SMBG according to FGM manufactures guideline and handling of trend arrows etc.
  Arms: C) Flash glucose monitoring (FGM); D) Carbohydrate counting, automated bolus calculation, FGM

SUMMARY:
This study aims to compare the effect of flash glucose monitoring (FGM) with traditional self-monitoring of blood glucose (SMBG) with or without carbohydrate counting and automated bolus calculation, in patients with type 1 diabetes and poor metabolic control.

The investigators will include in total 200 patients recruited from 5 clinical sites in the Capital Region of Copenhagen.

The patients will be randomized into four groups; A) Standard diabetes training, i.e. group training in in general diabetes health issues, B) Group training in carbohydrate counting and automated bolus calculation, the app MySugr will be taught and downloaded, C) Group training as in group A, and instructed to use FGM, D) Group training as in group B, and besides training in the use of the app MySugr, also instructed to use FGM.

All patients are followed for 26 weeks with 6 clinical visits, group training (1 visit) and 2 telephone consultations.

The primary outcome is time spent in normoglycemia.

ELIGIBILITY:
Inclusion criteria:

* Age >/= 18 years
* HbA1c > 53 mmol/mol
* Type 1 diabetes more than 1 year
* Treated with basal and bolus insulin. Basal insulin can be taken once or twice daily. The percentage basal/bolus insulin should as judged by the investigator cover the patient's real need for basal insulin - if he or she is not eating and taking bolus
* Patients may or may not have knowledge on carbohydrate counting
* Patients may or may not have any experience with continuous glucose monitoring or FGM
* Patients have a personal smart phone
* Patients attend the outpatient clinic in one of the five study sites included in the study

Exclusion criteria:

* Use of an automatic bolus calculator on a daily basis within the last three months
* Daily use of continuous glucose monitoring or FGM on a daily basis within the last three months
* Use of insulin pump
* Use of Neutral Protamine Hagedorn insulin as long acting insulin (Insulatard, Humulin Retard) within the last three months
* Pregnant, breastfeeding, plan to get pregnant
* Gastroparesis
* Severe diabetes complications including proliferative retinopathy and myocardial infarction within the last six months
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation as e.g. alcohol and drug abuse
* Current participation in another diabetes-related clinical trial that, in the judgment of the principle investigator, will compromise the results of the study or the safety of the subject
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Inability to understand the individual information and to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Time in normoglycemia | 26 weeks
  Difference in time in normoglycemic range 4-10 mmol/l at end of study measured by 2 weeks blinded FGM between group A (control group) and C (FGM) (min/day).

SECONDARY OUTCOMES:
HbA1c | 26 weeks
  Difference among groups in change in HbA1c (mmol/mol).
Severe hypoglycemia | 26 weeks
  Difference among groups in occurrence of severe hypoglycemia (defined as an event requiring assistance of another person. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal) (number of events during study period).
Hypoglycemia | 26 weeks
  Difference among groups in occurrence of symptomatic and confirmed hypoglycemia (< 3 mmol/l) (number of episodes per week).
Diabetes distress | 26 weeks
  Difference in changes in diabetes distress by the use of Problem Areas in Diabetes Questionnaire (PAID, score 0-100; higher scores reflecting diabetes distress).
Diabetes treatment satisfaction | 26 weeks
  Difference in changes in treatment satisfaction by the use of Diabetes Treatment Satisfaction Questionnaire (DTSQ, score 0-36; higher scores reflecting higher satisfaction).
Diabetes empowerment | 26 weeks
  Difference in changes in empowerment by the use of Diabetes empowerment test (DES-short form, containing 8 items, higher scores reflecting diabetes-related psychosocial self-efficacy. An item checked "strongly agree" receives 5 points; "agree" - 4 points; "neutral" - 3 points; "disagree" - 2 points; and "strongly disagree" receives 1 point, and an overall score is calculated by adding all of the scores (8-40) and dividing by the number of completed items (highest number is 8)).
Diabetes quality of life | 26 weeks
  Difference in changes in life quality by the use of Diabetes quality of life (ADDQoL-19, scores -9-3, lower scores reflecting maximum negative impact).
Blinded FGM hypoglycemia | 26 weeks
  Difference in change in time spent in hypoglycemia (<3mmol/l, <4 mmol/l) (min/day) from baseline (2 weeks) to end of study (2 weeks) in the different study groups.
Blinded FGM hyperglycemia | 26 weeks
  Difference in change in time spent in hyperglycemia (>10 mmol/l) (min/day) from baseline (2 weeks) to end of study (2 weeks) in the different study groups.
Blinded FGM glycemic variability | 26 weeks
  Difference in change in glycemic variability (standard deviation) from baseline (2 weeks) to end of study (2 weeks) in the different study groups.
Personality traits | 26 weeks
  Association between personality traits evaluated by the use of Neuroticism Extraversion Openness Agreeableness Conscientiousness Five-Factor Inventory-3 (NEO-Five Factors Inventory-3) questionnaire and any other outcome measures in the different groups. The NEO-Five Factors Inventory-3 covers five factors/domains that describe the commonly accepted personality traits. The inventory contains 60 statements that should be evaluated by self-ratings on a 5-point scale where 1 reflects "strongly disagree" and 5 reflects "strongly agree". The answers are related to the norm and based on these scores, personality traits are reported by the internet based Hogrefe Testsystem 5 (Hogrefe Publishing Group).
Total insulin dose | 26 weeks
  Difference in change between the groups in total insulin dose (units/day/kg) recorded as a mean of 2 weeks during FGM blinded measurements.
Total basal insulin dose | 26 weeks
  Difference in change between the groups in total basal insulin dose (units/day/kg) recorded as a mean of 2 weeks during FGM blinded measurements.
Insulin boluses | 26 weeks
  Difference in change between the groups in number of insulin boluses per day (number/day) recorded as a mean of 2 weeks during FGM blinded measurements.
Body weight | 26 weeks
  Difference among groups in body weight (kg).
Urinary albumin/excretion rate | 26 weeks
  Difference among groups in urinary albumin/excretion rate (mg/24 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Secher AL, Pedersen-Bjergaard U, Svendsen OL, Gade-Rasmussen B, Almdal T, Raimond L, Vistisen D, Norgaard K. Flash glucose monitoring and automated bolus calculation in type 1 diabetes treated with multiple daily insulin injections: a 26 week randomised, controlled, multicentre trial. Diabetologia. 2021 Dec;64(12):2713-2724. doi: 10.1007/s00125-021-05555-8. Epub 2021 Sep 8. PMID 34495375
- [Derived] Secher AL, Pedersen-Bjergaard U, Svendsen OL, Gade-Rasmussen B, Almdal TP, Dorflinger L, Vistisen D, Norgaard K. Study protocol for optimising glycaemic control in type 1 diabetes treated with multiple daily insulin injections: intermittently scanned continuous glucose monitoring, carbohydrate counting with automated bolus calculation, or both? A randomised controlled trial. BMJ Open. 2020 Apr 27;10(4):e036474. doi: 10.1136/bmjopen-2019-036474. PMID 32345699